CLINICAL TRIAL: NCT04210414
Title: Transfer of Single Embryo on Day 3 or 5 When Only One Embryo Transfer
Brief Title: Cleave-stage Transfer on Day 3 Versus Day 5 Transfer When Only One Embryo Available
Acronym: Cleave-blast
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID19 Pandemic affected recruitment across 2020 and the stringent inclusion criteria makes the proposed sample size to be likely unachievable in reasonable period.
Sponsor: Ibn Sina Hospital (Other Government)
Responsible Party: Principal Investigator, Muhammad Fawzy, IVF Lab Director, Ibn Sina Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: IbnSina-ET
Record Dates: First submitted 2019-12-21; First posted 2019-12-24 (Actual); Last update posted 2022-06-15 (Actual); Status verified 2022-06

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility | interventions — Embryo Transfer

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Day 3 transfer (Experimental): Transfer on day 3 when only one embryo is available
  Interventions: Other: Embryo transfer
- Day 5 transfer (Experimental): Transfer on day 5 when only one embryo is available
  Interventions: Other: Embryo transfer

INTERVENTIONS:
Other: Embryo transfer — Transfer of only one embryo

SUMMARY:
When only one embryo is available after in vitro fertilization, the option is to transfer either day 3 or day 5. There is no randomized trial compared the day 3 to day 5 for this subgroup.

DETAILED DESCRIPTION:
Recruitment is very slow. The TSC will discuss termination next meeting with the DMC.

ELIGIBILITY:
Inclusion Criteria:

* Infertile couple with only one embryo available for transfer

Exclusion Criteria:

* ineligible for study

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 83 (Actual)
Dates: Start 2020-01-10 (Actual); Primary Completion 2021-11-10 (Actual); Study Completion 2021-11-10 (Actual)

PRIMARY OUTCOMES:
Ongoing pregnancy rate | within 20 weeks of gestation

SECONDARY OUTCOMES:
Biochemical pregnancy rate | One month
clinical pregnancy | 7 weeks of gestation
Embryo development after In vitro fertilization cycle | 6 days after in vitro fertilization

CONTACTS AND LOCATIONS:
Locations (3):
- Egypt (3):
  - Qena Fertility Center, Qina, Qena Governorate
  - Banon Assiut, Asyut
  - IbnSina IVF Center, IbnSina Hospital, Sohag

IPD SHARING:
Plan to Share IPD: No